CLINICAL TRIAL: NCT06891911
Title: Groceries for Residents of Southeastern USA to Stop Hypertension
Acronym: GoFreshSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other); University of Vermont (Other)
Responsible Party: Principal Investigator, Stephen Juraschek, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P000102; GRT67144 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Elevated Blood Pressure; Cardiovascular Diseases; Dietary Intervention
Keywords: Hypertension; Dash Diet; Low Sodium; Diet; Nutrition; Clinical trial; Dietitian
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Individual, parallel, randomized control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The interventionists are masked to study outcomes. The participants and dietitian interventionists are masked to study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietitian-Assisted DASH Groceries (Experimental): Participants will order groceries sufficient to meet their caloric needs each week for 4 weeks with the assistance of a dietitian/nutrition interventionist. Groceries will be delivered to participants' homes or picked up at a convenient location. The dietitian/nutrition interventionist will provide brief educational content at the time of food delivery. Orders will be placed via phone or through virtual counseling sessions.
  Interventions: Behavioral: Dietitian-Assisted DASH groceries
- Self-directed shopping (Active Comparator): Participants will receive a stipend and some basic information about healthy eating. The stipend is not restricted to foods.
  Interventions: Behavioral: Self-directed shopping

INTERVENTIONS:
Behavioral: Dietitian-Assisted DASH groceries — The DASH ("Dietary Approaches to Stop Hypertension"), is a healthy dietary pattern that lowers blood pressure without reducing weight. The DASH diet emphasizes fruits, vegetables, and low-fat dairy products; includes whole grains, poultry, fish, and nuts; and is reduced in red meat, sweets, and sugar-containing beverages.
  Intervention Phase:
  This intervention is a weekly, 4-week DASH dietary intervention. A dietitian will assist participants in ordering groceries in a pattern consistent with the DASH diet to be delivered to their homes. The quantity of groceries will be based on participant Calorie needs and family size.
  Arms: Dietitian-Assisted DASH Groceries
Behavioral: Self-directed shopping — Intervention Phase:
  Participants will receive some basic information on healthy eating and a stipend during the 4-week intervention period. They are permitted to use the stipend however they choose and will not be asked about how they spent these funds.
  Arms: Self-directed shopping

SUMMARY:
GoFreshSE is a randomized control trial, testing the effects of a home-delivered, dietitian-assisted, DASH-patterned grocery intervention on blood pressure in adults with high blood pressure in Florida, Georgia, and Tennessee.

DETAILED DESCRIPTION:
Hypertension (HTN) affects half of US adults and is one of the most important modifiable risk factors for cardiovascular disease (CVD) and death.

The DASH diet is a proven strategy for lowering blood pressure in adults. Our proposed clinical trial will evaluate the effectiveness of a scalable solution: home-delivered, low-sodium groceries aligned with the DASH dietary pattern and ordered with dietitian assistance via a virtual supermarket, in reducing blood pressure.

Participants will be assigned to one of two 1-month long interventions: (1) dietitian-assisted, DASH-patterned, home-delivered groceries ordered weekly through Amazon Fresh (or Whole Foods) over 4 weeks or (2) self-directed grocery shopping (monthly stipend and DASH diet brochure) (referent).

ELIGIBILITY:
Inclusion Criteria:

1. Resting systolic blood pressure of 120 to <160 mm Hg and diastolic blood pressure <110 mm Hg
2. Resident of Florida, Georgia, and Tennessee
3. Able to receive home-delivered groceries or pick them up at a convenient location and willing to eat only the groceries provided over a 4-week period
4. Have access to refrigeration, cooking appliances, and Wi-Fi/cellular service
5. Have access to mobile device or computer to be able to conduct grocery orders via video conference and send/receive text messages
6. Willing and able to complete required measurement procedures
7. Able to provide consent for the study
8. Has access to a primary care team, urgent care center, or emergency room the study team can refer to for follow up care if warranted during the study

Exclusion Criteria:

A. Laboratory Exclusions:

1. Serum potassium ≥5.0 mmol/L or <3.5 mmol/L
2. Estimated glomerular filtration rate (eGFR) <30 mL/min per 1.73 m^2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
3. Hemoglobin A1c ≥6.5%

B. Medication Exclusions:

Unstable doses (i.e. a change in the 6 months prior to screening or randomization or planning to start within study period) of the following:

1. GLP-1 and dual GLP-1/GIP receptor agonists
2. Anti-hypertension medications
3. Sodium-glucose co-transporter 2 (SGLT2) inhibitors
4. Glucose lowering medications

Use of any of the following medications:

1. Potassium supplement, except if part of a multivitamin
2. Warfarin (Coumadin)
3. Chronic oral corticosteroid (intermittent use is okay)
4. Weight loss medications (non-GLP-1 receptor agonists)
5. Sulfonylurea or any insulin use

Any medication not compatible with participation as determined by the investigators

C. Physical Exclusions:

1. Systolic blood pressure: <120 or ≥160 mm Hg or diastolic blood pressure ≥110 mm Hg
2. Arm circumference >52 cm (or the upper limit of the validated BP device)

D. Medical History Exclusions:

1. Self-reported weight loss or gain of 15 pounds during prior 2 months
2. Active cardiovascular disease or any event in the prior 6 months, including coronary artery bypass grafting (CABG), percutaneous transluminal coronary angioplasty (PTCA), myocardial infarction (MI), cerebrovascular accident (CVA), or congestive heart failure (CHF) exacerbation requiring hospital admission
3. Cancer diagnosis or treatment in the last 2 years (non-melanoma skin cancer or localized breast or prostate or bladder cancer not requiring systemic therapy is acceptable)
4. Gastrointestinal surgery or history that affects nutrition absorption or requires a specific diet that will deter DASH diet adherence
5. Pregnancy or lactation or planned pregnancy during the study period
6. Any emergency department (ED) visit for asthma or chronic obstructive pulmonary disease (COPD) in the last 6 months
7. Hypoglycemia hospitalization in the last 12 months
8. Any other serious illness or condition not compatible with participation as determined by the investigators

E. Lifestyle and Other Exclusions:

1. Significant food allergies, preferences, intolerances, or dietary requirements that would interfere with diet adherence
2. Consumption of more than 14 alcoholic drinks per week or consumption of more than 6 drinks on one or more occasion per week
3. Active substance use disorder that would interfere with participation
4. Extreme food insecurity
5. Participation in or planning to start weight loss program
6. Current participation in another clinical trial that could interfere with the study protocol
7. Anticipated change in residence outside of eligible states prior to the end of the study
8. Families with more than 6 adults at dinner time (children count as half an adult)

F. Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Self-measured systolic blood pressure | Measured before and after the 4-week intervention
  This entails 4 measurements, 2 in the morning and 2 in the evening, over a 7 day period (at least 3 concurrent days is acceptable for analysis).

SECONDARY OUTCOMES:
Self-measured diastolic blood pressure | Measured before and after the 4-week intervention
  This entails 4 measurements, 2 in the morning and 2 in the evening, over a 7 day period (at least 3 concurrent days is acceptable for analysis).
Seated systolic and diastolic blood pressure (technician-measured) | Measured before and after the 4-week intervention
  Seated systolic and diastolic blood pressure measured by a technician in participants' homes, using the office blood pressure device.
Body Mass Index (BMI) | Height is measured before the intervention. Weight is measured before and after the 4-week intervention.
  At home measurement based on height and weight measured by a technician via a stadiometer and scale.
24-hour dietary recall | Measured before and after the 4-week intervention
  Assessed via self-administered questionnaire using the Automated Self-Administered 24-Hour Dietary Recall (ASA24).
Spot urine sodium/potassium ratio | Measured before and after the 4-week intervention
  Measured in urine collected at the participants' homes.
Lipids | Measured before and after the 4-week intervention
  Measured in fasted serum specimens collected during phlebotomy. Includes total cholesterol, high density lipoprotein cholesterol, derived low density lipoprotein cholesterol, and triglycerides
Fasting glucose | Measured before and after the 4-week intervention
  Measured in blood as part of a basic metabolic panel
Serum potassium | Measured before and after the 4-week intervention
  Measured in blood as part of a basic metabolic panel

OTHER OUTCOMES:
General Health Status | Measured before and after the 4-week intervention
  Single General Health Status Question: "Would you say that in general your health is excellent, very good, good, fair, or poor?"
Financial strain | Measured before and after the 4-week intervention
  We will ask the following questions: How often does this describe you? I don't have money to pay my bills (including food, housing, medical care or heating).
  Never / Rarely / Sometimes / Often / Always

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP